CLINICAL TRIAL: NCT02085278
Title: Safety of Apollo Embolization Delivery Micro Catheter in Pediatric Patients With Vascular Malformations
Brief Title: Safety of Apollo Micro Catheter in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: APL01
Record Dates: First submitted 2014-03-04; First posted 2014-03-12 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Brain Arteriovenous Malformation; Brain Vascular Malformations; Vein of Galen Malformation
Keywords: arteriovenous malformation; Brain; AVM; Onyx; Micro catheter; catheter entrapment,; Embolization; Vein Of Galen
MeSH Terms: conditions — Central Nervous System Vascular Malformations; Vein of Galen Malformations; Arteriovenous Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apollo Group (Experimental): Apollo Micro catheter device
  Interventions: Device: Apollo Micro Catheter device

INTERVENTIONS:
Device: Apollo Micro Catheter device — Detachable Tip Micro catheter

SUMMARY:
This is a clinical trial/study for patients diagnosed with brain arteriovenous malformation (AVM). An AVM is an abnormal connection between the arteries and veins of the brain. Patients considered for this trial are 21 years and younger with AVM suitable for embolization treatment (a procedure used to block the abnormal connection between the arteries and veins of the brain) with Onyx Liquid Embolic System (Onyx LES) or TruFill n-Butyl Cyanoacrylate (n-BCA) Liquid Embolic System (both are liquid substances used in the embolization procedure to block the abnormal connection).

DETAILED DESCRIPTION:
-Why is this study being done?

The purpose of this study is to evaluate the safety of the Apollo Embolization Delivery Micro Catheter device (device that looks like a long thin hallow tube) when used in Pediatric patients with vascular malformations.

The Apollo Onyx Delivery Micro Catheter device is manufactured by Micro Therapeutics, Inc. d/b/a ev3 Neurovascular. Apollo Onyx™ Delivery Micro Catheter device is not approved for use in the U.S, although it is widely used and approved for use in Europe (CE0297).

This clinical study is sponsored by Dr. Alejandro Berenstein of St.Luke's-Roosevelt Hospital, New York who is also the principal Investigator of the study. Total duration of study is up to 30 months with approximately an 18 months enrollment period. Patients follow up period is up to 12 months upon enrollment.

ELIGIBILITY:
Inclusion Criteria:

* The subject or subject's legally authorized representative has signed and dated an informed Consent Form.
* Subject's age is ≤ 21 years.
* The subject has a confirmed diagnosis of brain arteriovenous malformation in the cerebral cortex, cerebellum or dura mater that is indicated for endovascular embolization with Onyx™ LES or TruFill n-Butyl Cyanoacrylate (n-BCA) Liquid Embolic Systems and where the use of Apollo Embolization Delivery Micro Catheter may or may not be indicated for surgical resection.
* The subject is clinically and neurologically stable for a minimum of 48 hours prior to embolization.
* The subject has a life expectancy of at least 1 year with the exception of new born babies with Vein of Galen malformation with cardiopulmonary failure where no other treatment option remains.
* The subject agrees to and is capable of completing all study required procedures

Exclusion Criteria:

* Female who is pregnant or lactating.
* Current participation in another investigational drug or device study.
* Subject has a brain tumor or other malignancy

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The study's primary endpoint is the incidence of catheter entrapment. | Within 24 hours after embolization
  The study's primary endpoint is the incidence of catheter entrapment. Catheter entrapment entails any part of the Apollo Micro catheter Delivery Device, excluding the catheter tip, being inadvertently left within the vasculature at the end of the procedure

SECONDARY OUTCOMES:
Incidence of unintentional catheter tip detachment. | Within 24 hours after embolization
  Defined by the separation of the detachment joint during the procedure either during navigation, prior to embolization completion, or upon catheter retrieval when distal tip is not entrapped in Onyx cast.
Incidence of migration of the detached catheter tip. | Within 24 hours after embolization
  Defined by an observed change in position of the detached tip during post embolization imaging.
Incidence of catheter/procedure-related adverse events. | At one year post procedure
  The adverse events include but not limited to vascular occlusion (a sudden blockage of a blood vessel usually with a blood clot), vascular thrombosis (acute and subacute) (blood clots in a vessel that break loose and enter another vessel), allergic reactions, thrombocytopenia (significant decrease in red blood cell clotting factors), Death, neurologic deterioration (nervous system decline) including stroke and death, pulmonary embolization or complications (blockage of blood vessels in the lung), perforation or dissection of the vessel (tear of the blood vessel).
Incidence of catheter/tip leakage from the detachment zone. | At one year post procedure
Incidence of migration of the detached catheter tip | At one year post procedure
  Defined by an observed change in position of the detached tip during the post embolization imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Otokiti, MBBS, Study Director — St. Luke's-Roosevelt Hospital Center; Alejandro Berenstein, M.D, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (1):
- St.Luke's-Roosevelt Hospital, New York, New York, United States

REFERENCES:
- [Background] Chang SD, Marcellus ML, Marks MP, Levy RP, Do HM, Steinberg GK. Multimodality treatment of giant intracranial arteriovenous malformations. Neurosurgery. 2003 Jul;53(1):1-11; discussion 11-3. doi: 10.1227/01.neu.0000068700.68238.84. PMID 12823868
- [Background] Walcott BP, Gerrard JL, Nogueira RG, Nahed BV, Terry AR, Ogilvy CS. Microsurgical retrieval of an endovascular microcatheter trapped during Onyx embolization of a cerebral arteriovenous malformation. J Neurointerv Surg. 2011 Mar;3(1):77-9. doi: 10.1136/jnis.2010.002733. Epub 2010 Oct 5. PMID 21990795
- [Background] Santillan A, Zink W, Knopman J, Riina H, Gobin YP. Balloon-assisted technique for trapped microcatheter retrieval following onyx embolization. A case report. Interv Neuroradiol. 2009 Dec;15(4):453-5. doi: 10.1177/159101990901500414. Epub 2009 Dec 28. PMID 20465885
- [Background] Newman CB, Park MS, Kerber CW, Levy ML, Barr JD, Pakbaz RS. Over-the-catheter retrieval of a retained microcatheter following Onyx embolization: a technical report. J Neurointerv Surg. 2012 Jul;4(4):e13. doi: 10.1136/neurintsurg-2011-010040. Epub 2011 Jun 16. PMID 21990504